CLINICAL TRIAL: NCT04791683
Title: The Effect of Sexual Counseling Given to Infertile Couples in Line With PLISSIT Model on Sexual Function and Sexual Satisfaction
Brief Title: Sexual Counseling According to the PLISSIT Model in Primary Infertile Couples
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ezgi SAHİN, Msc, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 13022260-300-108795
Record Dates: First submitted 2021-03-07; First posted 2021-03-10 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Infertility; Sexuality; Sexual Dysfunction; Nurse's Role; Infertility; Female; Infertility, Male
MeSH Terms: conditions — Infertility; Sexuality; Sexual Dysfunction, Physiological; Infertility, Female; Infertility, Male

STUDY DESIGN:
Intervention Model Description: Parallel assignment Randomized controlled experimental study
Who Masked: Participant
Masking Description: Single (Participant) In the single-blind method,subjects do not know which of the experimental or control goups they were selected and therefore which method was applied to them. The researcher konows the subjects selected for the experimental and control groups, and therefore which method was applied to which subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Infertile couples in the control group were selected by randomization, routine protocols in the clinic were applied
- Experimental (Experimental): 1. st interview: Application of data collection tools
  2. nd meeting: Sexual counseling (1 week after the first interview)
  3. rd interview: Sexual counseling (1 week after the first session)
  4. th meeting: Sexual counseling (1 week after the second session)
  5. th interview: Telephone interview (2 months after the first assessment)
  6. th interview: re-application of data collection tools, including the final evaluation
  Interventions: Other: sexaul counseling

INTERVENTIONS:
Other: sexaul counseling — Sexual counseling includes interviews about sexual problems in couples who are in the process of infertility treatment and suggestions for solving these problems.
  Arms: Experimental

SUMMARY:
This study was planned to determine the effect of sexual counseling given to primary infertile couples in line with the PLISSIT model on sexual function and sexual satisfaction.

DETAILED DESCRIPTION:
The study will be conducted in the Infertility clinic of a medical faculty hospital. Couples receiving primary infertility treatment will be included in the study. It is planned to apply "Introductory Information Form, Female Sexual Function Index, Arizona Sexual Experiences Scale Male Form, Beck Depression Scale, New Sexual Satisfaction Scale and Infertility Stress Scale" to the experimental and control groups in the pre-initial evaluation. Within the scope of sexual counseling to be given to the couples in the experimental group in line with the PLISSIT Model; In order to increase the level of sexual function and sexual satisfaction, education of reproductive system anatomy and physiology, providing information about how the infertility process and treatment can affect sexual functions, determining the problems related to sexual health, trying to eliminate the misinformation and myths about sexuality, It is planned to include suggestions such as helping to cope well, alternative sexual intercourse positions according to the needs of the couples, body exploring exercise, sexual organs exploration exercise, masturbation exercise, kegel exercise.

The experimental group will be given an appointment for "sexual counseling" sessions held in 3 sessions at least 1 week apart. Each of these sessions will be completed in 60 minutes. Before the interviews, in line with the literature, "Sexual Counseling Booklet for Infertile Couples" will be prepared. In line with the scope of sexual counseling, the study is planned to be terminated by conducting 5 face-to-face interviews and 1 phone call with the experimental group. In the final evaluation, in order to determine the effects of sexual counseling on sexual health with the experimental group, the 'Introductory Information Form', Female Sexual Function Index, Male Form of Arizona Sexual Experiences Scale, New Sexual Satisfaction Scale and Infertility Stress Scale, at the appointment dates planned on the 3rd month after the first interview. '' The research will be terminated by filling in a face-to-face interview.

The couples in the control group will be interviewed in the second month after the first interview, and on the appointment dates scheduled for the 3rd month after the first interview, '' Introductory Information Form, Female Sexual Function Index, Arizona Sexual Experiences Scale Male Form, New Sexual Satisfaction Scale. and Infertility Stress Scale '' will be filled again with a face-to-face interview, and the research will be terminated.

ELIGIBILITY:
Inclusion Criteria:

* Sexual dysfunction in infertile men and women (FSFI = 26.55 points and below, ---ASEX≥11 points and above)
* Having been diagnosed with infertility at least a year ago
* Being in the diagnostic test phase
* On the day of vaccination
* After IVF / ICSI-Embryo Transfer
* 18-45 years of age
* Being literate,

Exclusion Criteria:

* Having a chronic disease other than infertility
* With a psychiatric illness
* Have any chronic disease
* Couples with Secondary Infertility
* IVF / ICSI-OPU (Egg pick up)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — men and women receiving infertility treatment
Enrollment: 60 (Estimated)
Dates: Start 2019-08-19 (Actual); Primary Completion 2021-04-20 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
The Female Sexual Function Index | The first assessment (ie first measurements) of sexual function levels is made on the first day of diagnostic tests for both groups of women attending the infertility clinic.
  The levels of desire, arousal, lubrication, orgasm, satisfaction and sexual pain in women are evaluated in the first and final evaluation
The Female Sexual Function Index | The final assessment of sexual function levels (ie the last measurements) is made for women in both groups, on average 12 weeks after the initial assessment.
  The levels of desire, arousal, lubrication, orgasm, satisfaction and sexual pain in women are evaluated in the first and final evaluation
Arizona Sexual Experiences Scale Male Form | The first assessment (ie first measurements) of sexual function levels is made on the first day of diagnostic tests for both groups of men attending the infertility clinic.
  In the first evaluation and in the final evaluation, the sexual function level of men and the sexual problems that arise are evaluated.
Arizona Sexual Experiences Scale Male Form | The final assessment of sexual function levels (ie the last measurements) is made for men in both groups, on average 12 weeks after the initial assessment.
  In the first evaluation and in the final evaluation, the sexual function level of men and the sexual problems that arise are evaluated.
The New Sexual Satisfaction Scale | The first assessment of sexual satisfaction levels (ie the first measurements) is made on the first day of diagnostic tests for both male and female groups admitted to the infertility clinic.
  In the first and final evaluation, the self-centered sub-dimension, which is the first sub-dimension of the scale, measures the level of sexual satisfaction consisting mostly of personal experiences, while in the second sub-dimension, the co-partner / sexual activity-centered sub-dimension, the sexual behavior and reactions of the person's partner and also the diversity of sexual activity and / or the level of sexual satisfaction obtained from the frequency is evaluated.
The New Sexual Satisfaction Scale | The final assessment of sexual satisfaction levels (ie the last measurements) is made for men and women in both groups, on average, 12 weeks after the initial assessment.
  In the first and final evaluation, the self-centered sub-dimension, which is the first sub-dimension of the scale, measures the level of sexual satisfaction consisting mostly of personal experiences, while in the second sub-dimension, the co-partner / sexual activity-centered sub-dimension, the sexual behavior and reactions of the person's partner and also the diversity of sexual activity and / or the level of sexual satisfaction obtained from the frequency is evaluated.
Infertility Stress Scale | The first assessment of infertility stress levels (ie the first measurements) is made on the first day of diagnostic tests for both male and female groups attending the infertility clinic.
  In the first and last evaluation, stress in the personal sphere, stress in the marital sphere and stress in the social sphere are measured using the Infertility Stress Scale (ISI).
Infertility Stress Scale | The final assessment of infertility stress levels (ie final measurements) is made for men and women in both groups, on average 12 weeks after the initial assessment.
  In the first and last evaluation, stress in the personal sphere, stress in the marital sphere and stress in the social sphere are measured using the Infertility Stress Scale (ISI).
Beck Depression Inventory | The first assessment of depression levels (ie first measurements) is made on the first day of diagnostic tests for both male and female groups attending the infertility clinic.
  In the first evaluation, various symptoms and severity of depression that may exist in individuals are evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Ezgi ŞAHİN, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benksim A, Elkhoudri N, Addi RA, Baali A, Cherkaoui M. Difference between Primary and Secondary Infertility in Morocco: Frequencies and Associated Factors. Int J Fertil Steril. 2018 Jul;12(2):142-146. doi: 10.22074/ijfs.2018.5188. Epub 2018 Mar 18. PMID 29707931
- [Background] Brassard A, Dupuy E, Bergeron S, Shaver PR. Attachment insecurities and women's sexual function and satisfaction: the mediating roles of sexual self-esteem, sexual anxiety, and sexual assertiveness. J Sex Res. 2015;52(1):110-9. doi: 10.1080/00224499.2013.838744. Epub 2013 Dec 18. PMID 24350570
- [Background] Czyzkowska A, Awruk K, Janowski K. Sexual Satisfaction and Sexual Reactivity in Infertile Women: The Contribution of The Dyadic Functioning and Clinical Variables. Int J Fertil Steril. 2016 Jan-Mar;9(4):465-76. doi: 10.22074/ijfs.2015.4604. Epub 2015 Dec 23. PMID 26985333
- [Background] Farnam F, Janghorbani M, Raisi F, Merghati-Khoei E. Compare the effectiveness of PLISSIT and sexual health models on women's sexual problems in Tehran, Iran: a randomized controlled trial. J Sex Med. 2014 Nov;11(11):2679-89. doi: 10.1111/jsm.12659. Epub 2014 Aug 5. PMID 25091932
- [Background] Ferraresi SR, Lara LA, de Sa MF, Reis RM, Rosa e Silva AC. Current research on how infertility affects the sexuality of men and women. Recent Pat Endocr Metab Immune Drug Discov. 2013 Sep;7(3):198-202. doi: 10.2174/18722148113079990009. PMID 23829396
- [Background] Khakbazan Z, Daneshfar F, Behboodi-Moghadam Z, Nabavi SM, Ghasemzadeh S, Mehran A. The effectiveness of the Permission, Limited Information, Specific suggestions, Intensive Therapy (PLISSIT) model based sexual counseling on the sexual function of women with Multiple Sclerosis who are sexually active. Mult Scler Relat Disord. 2016 Jul;8:113-9. doi: 10.1016/j.msard.2016.05.007. Epub 2016 May 24. PMID 27456885